CLINICAL TRIAL: NCT05522361
Title: Risdiplam Exchange in Patients With Spinal Muscular Atrophy (SMA) Previously and Exclusively Treated With Nusinersen
Brief Title: Risdiplam in Patients With Spinal Muscular Atrophy Previously Treated With Nusinersen
Acronym: RISE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Clinic for Special Children (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kevin A. Strauss, MD, Medical Director, Clinic for Special Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISE
Record Dates: First submitted 2022-05-24; First posted 2022-08-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: nusinersen; prospective; risdiplam
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label crossover (Experimental): Participants crossover to 36 months of open-label risdiplam mono therapy following a comparable period of nusinersen treatment.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — administered to participants per product label insert

SUMMARY:
Risdiplam Exchange (RISE) is a study of spinal muscular atrophy (SMA) patients who crossover to 36 months of open-label risdiplam monotherapy following a comparable period of nusinersen treatment. The schedule of assessments (SOAs) carry over seamlessly for the cohort from studies done while treated with nusinersen and continue to track the most informative outcomes from that trial (e.g. nine hole peg test and grip strength), while adding the Box and Block Test (BBT) as an additional measure of upper limb endurance and function.

DETAILED DESCRIPTION:
Risdiplam is an orally bioavailable small molecule that distributes into the central nervous system (CNS) and peripheral tissues where it modifies SMN2 pre-mRNA splicing and increases tissue SMN protein levels. It was approved by the U.S. Food and Drug Administration for all SMA patients older than 2 months of age in August 2020.

Clinical trial data prompted us to consider risdiplam a reasonable alternative to nusinersen administered intrathecally or by subcutaneous intrathecal catheter (SIC) for patients with more advanced SMA. Considered within this clinical context, risdiplam presents a significant advantage by eliminating the risks of mechanical failure, intrathecal bleeding, and CNS infection associated with the SIC device. The schedule of assessments (SOAs) used in this cohort during the previous three-year period as part of a nusinersen study provide us with an established framework for data collection. Thus, the overall clinical experience with risdiplam as compared to nusinersen can be assessed using a prospective, crossover design in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Biallelic SMN1 deletions
* 3 or 4 copies of SMN2
* Prior treatment with nusinersen for a minimum of 22 months

Exclusion Criteria:

* Prior treatment with SMN gene replacement therapy
* Prior exposure to another investigational agent.
* Confounding neuromuscular disorder other than SMA

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Comparative intrasubject performance on nine hole peg test (NHPT) | 36 months
  Time in seconds to place and subsequently remove nine one inch pegs in holes assessed in dominant and non dominant hands

SECONDARY OUTCOMES:
Intrasubject changes in lower limb and overall motor function | 36 months
  Revised Hammersmith Scale (RHS) of 33 items with grades of 0 (unable),1 (attempted, not completed) and 2 (achieves task); the greater the sum total, the higher overall motor function.
Intrasubject changes in upper limb motor function | 36 months
  box and block test (BBT): number of 1 inch wood blocks moved from one compartment to an adjacent one over a wall within 5 minutes, with more blocks moved corresponding to higher upper limb motor function
Intrasubject change in pulmonary function | 36 months
  maximal inspiratory pressure (MIP) and mean expiratory pressure (MEP), measured in centimeters of water displaced
Frequency and type of adverse events | 36 months
  laboratory testing, self-reported, and observed during the study
Comparative intrasubject change in grip strength | 36 months
  hand-held dynamometry (MyoGrip and MyoPinch) measures force in Newtons

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Special Children, Strasburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strauss KA, Carson VJ, Brigatti KW, Young M, Robinson DL, Hendrickson C, Fox MD, Reed RM, Puffenberger EG, Mackenzie W, Miller F. Preliminary Safety and Tolerability of a Novel Subcutaneous Intrathecal Catheter System for Repeated Outpatient Dosing of Nusinersen to Children and Adults With Spinal Muscular Atrophy. J Pediatr Orthop. 2018 Nov/Dec;38(10):e610-e617. doi: 10.1097/BPO.0000000000001247. PMID 30134351
- [Background] Carson VJ, Young M, Brigatti KW, Robinson DL, Reed RM, Sohn J, Petrillo M, Farwell W, Miller F, Strauss KA. Nusinersen by subcutaneous intrathecal catheter for symptomatic spinal muscular atrophy patients with complex spine anatomy. Muscle Nerve. 2022 Jan;65(1):51-59. doi: 10.1002/mus.27425. Epub 2021 Oct 19. PMID 34606118
- [Background] Ribero VA, Daigl M, Marti Y, Gorni K, Evans R, Scott DA, Mahajan A, Abrams KR, Hawkins N. How does risdiplam compare with other treatments for Types 1-3 spinal muscular atrophy: a systematic literature review and indirect treatment comparison. J Comp Eff Res. 2022 Apr;11(5):347-370. doi: 10.2217/cer-2021-0216. Epub 2022 Jan 18. PMID 35040693